CLINICAL TRIAL: NCT05725018
Title: A Phase 3b Study for the Treatment of Dystrophic Epidermolysis Bullosa (DEB) in New and Previously EB-101 Treated Patients
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Abeona Therapeutics, Inc (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EB-101-CL-302
Record Dates: First submitted 2023-01-23; First posted 2023-02-13 (Actual); Last update posted 2025-06-27 (Actual); Status verified 2025-06

CONDITIONS: Epidermolysis Bullosa; Recessive Dystrophic Epidermolysis Bullosa; RDEB
Keywords: Chronic wounds
MeSH Terms: conditions — Epidermolysis Bullosa; Epidermolysis Bullosa Dystrophica

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- EB-101 Surgical application of RDEB wounds (Experimental): New or Previously Treated RDEB Patients
  Interventions: Biological: EB-101 Surgical application of RDEB wounds

INTERVENTIONS:
Biological: EB-101 Surgical application of RDEB wounds — EB-101 autologous RDEB keratinocytes isolated from skin biopsies and transduced with a recombinant retrovirus containing a full-length COL7A1 expression cassette for C7
  Other Names:
  • LZRSE-Col7A1 Engineered Autologous Epidermal Sheets [LEAES]
  Other Names: pz-cel

SUMMARY:
To evaluate and further characterize the safety of EB-101 (LZRSE-Col7A1 gene-corrected keratinocyte sheets with type VII collagen [C7] expression) for the treatment of large, chronic DEB wounds in new and previously EB-101 treated patients 12 months and older.

DETAILED DESCRIPTION:
A multicenter, open-label, single-arm Phase 3b safety study of one-time surgical application of up to 12 autologous, LZRSE-Col7A1 gene-corrected keratinocyte sheets with C7 expression (EB-101) for the treatment of large, chronic DEB wounds in each of approximately 10-12 patients. Patients enrolled will also contribute biopsies to support manufacturing requirements. All patients will be followed through 24 weeks post-treatment.

Patients will be evaluated at their Screening Visit (D -60 to D -25), a phone call approximately 14 days after screening, and at Baseline (Day -1) prior to treatment on Day 0. Patients will remain in the hospital, or other suitable inpatient medical facility that will allow appropriate immobilization of treated wounds, as determined by the Investigator, for observation for up to 7 days (±2 days) following treatment. They will be evaluated by phone on Day 14; by telehealth visits on Weeks 4, 8, and 18; and by clinic visits on Weeks 12 and 24.

ELIGIBILITY:
Inclusion Criteria:

1. Clinical diagnosis of DEB.
2. Age 12 months and older.
3. Willing and able to give consent/assent; if under the age of 18 years, guardian(s) is/are willing and able to give consent.
4. (This inclusion criterion was deleted as of Amendment 1.)
5. Confirmation of DEB diagnosis (either dominant [DDEB] or recessive [RDEB] forms) by genetic testing.
6. Able to undergo adequate anesthesia during EB-101 treatment.
7. All women of childbearing potential must have a negative urine pregnancy test and use a reliable birth control method throughout the duration of the study.
8. On stable pain medication regimen for at least 30 days prior to Screening (and through Baseline).
9. Must have at least one wound site that meets all of the following criteria:

   1. An area ≥20 cm2,
   2. Present for ≥6 months, and
   3. Stage 2 wound defined as an open skin wound with partial thickness loss of dermis that has not extended through the dermis into subcutaneous tissue.
10. For patients with RDEB, they must have had Vyjuvek exposure by the time of screening or positive anti-C7 antibodies at baseline.
11. Patients must be willing to discontinue Vyjuvek and Filsuvez use on EB-101 treated sites until completion of the Week 24 visit.

Exclusion Criteria:

1. Medical instability limiting ability to travel to the study site or undergo EB-101 treatment.
2. The presence of medical illness expected to complicate participation and/or compromise the safety of this technique, such as active infection with human immunodeficiency virus (HIV), hepatitis B, or hepatitis C.
3. (This exclusion criterion was deleted as of Amendment 3.)
4. Evidence of systemic infection.
5. Current evidence or a history of SCC in the area that will undergo EB-101 application.
6. Active drug or alcohol addiction.
7. Hypersensitivity to vancomycin or amikacin.
8. Receipt of chemical or biological investigational therapy for the specific treatment of DEB in the 3 months prior to EB-101 application.
9. Breast-feeding.
10. Inability to properly follow protocol assessments and protect keratinocyte sheet sites as determined by the PI.
11. Grade 3 clinical event or laboratory abnormality at Day 0. Abnormalities such as esophageal strictures, anemia, low albumin, and pain/itch are expected in severe DEB patients, and these abnormalities will not exclude a patient.
12. Unwillingness or inability to provide 4 skin biopsies, or patient's keratinocytes cannot be manufactured for use in EB-101 application.
13. Any other circumstance where the PI believes that the patient may not be appropriate for participation in the study.

Min Age: 12 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2023-04-02 (Actual); Primary Completion 2025-09-30 (Estimated); Study Completion 2025-09-30 (Estimated)

PRIMARY OUTCOMES:
Safety Endpoint (number of treatment-related and treatment-emergent adverse events (AEs) and serious adverse events (SAEs) | 6 months
  The number of treatment-related and treatment-emergent adverse events (TEAEs), treatment-emergent wound adverse events (TEWAEs), and serious adverse events (SAEs), including systemic and wound-specific adverse events.
Safety Endpoint (number of patients and wounds that have an infection or any related adverse event.) | 6 months
  The number of patients and wounds that have an infection or any related adverse event (AE).
Safety Endpoint (number of patients and wounds that result in hospitalization (serious adverse event ) | 6 months
  The number of patients and wounds that result in hospitalization (SAE).
Safety Endpoint (Incidence of squamous cell carcinoma) | 6 months
  The incidence of squamous cell carcinoma (SCC).
Safety Endpoint RCR status | 6 months
  Replication-competent retrovirus (RCR) status.

OTHER OUTCOMES:
Proportion of RDEB wounds with ≥50%, ≥75%, and complete | 6 months
  Proportion of RDEB wounds with ≥50%, ≥75%, and complete (i.e., re epithelialization with no drainage or erosion and presence of only minor crusting) healing at Weeks 12 and 24, as determined by direct Investigator assessment.
Extent of pain reduction assessed by the Wong-Baker FACES scale | 6 months
  Extent of pain reduction assessed by the Wong-Baker FACES scale (for patients ages ≥6 years old) at Weeks 8, 12, and 24.
Longitudinal change in scores of Worst Itch Numeric Rating Scale | 6 months
  Longitudinal change in scores of Worst Itch Numeric Rating Scale (WI-NRS; for patients ages ≥6 years old) scores assessed at Weeks 8, 12, and 24
Longitudinal change of Zarit Burden Interview Short Form | 6 months
  Longitudinal change of Zarit Burden Interview Short Form (ZBI-12) for caregiver scores related to wound care, assessed at Weeks 12 and 24 (for all ages).
Change in Quality of Life in Epidermolysis Bullosa | 6 months
  Change in Quality of Life in Epidermolysis Bullosa (QOLEB) scores assessed at Week 24 compared with pretreatment Baseline scores (completed by patients ≥11 years old or with guidance for patients 8 to 10 years old). If patient is <8 years old, QOLEB should be completed by a legal guardian.
Change in Caregiver Global Impression of Pain | 6 months
  Change in Caregiver Global Impression of Pain (CrGI-Pain) scores assessed at Weeks 8, 12, and 24 compared with pretreatment Baseline (for all ages).
Comparison of how non-collagenous region 1 of the collagen VII molecule | 6 months
  Comparison of how non-collagenous region 1 of the collagen VII molecule (NC1) status relates to wound healing and safety profile (if applicable).
Comparison of how circulating C7 antibody status relates to wound healing and safety profile | 6 months
  Comparison of how circulating C7 antibody status relates to wound healing and safety profile (if applicable).

CONTACTS AND LOCATIONS:
Overall Officials: Angela Iheanacho, MS, Study Director — Abeona Therapeutics, Inc; Sarah Abdelwahab, MD, Study Director — Abeona Therapeutics, Inc
Locations (2):
- United States (2):
  - Stanford University, Redwood City, California
  - University of Massachusetts Medical School, Worcester, Massachusetts

IPD SHARING:
Plan to Share IPD: No